CLINICAL TRIAL: NCT03006445
Title: Official Title: Safety and Efficacy Evaluation Study of FYU-981 Long-term Administration for Hyperuricemia With or Without Gout (Phase III Study)
Brief Title: Study of FYU-981 in Hyperuricemia With or Without Gout
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fuji Yakuhin Co., Ltd. (Industry)
Collaborators: Mochida Pharmaceutical Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FYU-981-010
Record Dates: First submitted 2016-12-28; First posted 2016-12-30 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2017-09

CONDITIONS: Hyperuricemia With or Without Gout
MeSH Terms: interventions — dotinurad

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FYU-981 (Experimental)
  Interventions: Drug: FYU-981

INTERVENTIONS:
Drug: FYU-981

SUMMARY:
The purpose of this study is confirmatory investigation of safety and efficacy of FYU-981 administered orally to hyperuricemic patients with and without gout for 34 or 58 weeks by the method of multicenter, open label and ascending dose regimen.

ELIGIBILITY:
Inclusion Criteria:

* Hyperuricemic or gout patients
* Serum urate level:

>= 7.0mg/dL in patients with history of gout, or >= 8.0mg/dL in patients with hypertension, diabetes or metabolic syndrome, or >= 9.0mg/dL

Exclusion Criteria:

* Gouty arthritis within two weeks before start of study treatment
* Secondary hyperuricemia
* HbA1c: >= 8.4%
* Uric acid-overproduction type in the classification of hyperuricemia
* History of, clinically significant cardiac, hematologic and hepatic disease
* Kidney calculi or clinically significant urinary calculi
* eGFR: < 30mL/min/1.73m^2
* Systolic blood pressure: >= 180 mmHg
* Diastolic blood pressure: >= 110 mmHg

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Percent reduction from baseline in serum urate level at the final visit | 34 or 58 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan

REFERENCES:
- [Derived] Takahashi T, Beppu T, Hosoya T, Yokota N. Changes in urinary albumin levels with dotinurad oral administration in hyperuricemic patients with microalbuminuria: a post hoc analysis. Clin Exp Nephrol. 2025 Oct;29(10):1384-1393. doi: 10.1007/s10157-025-02750-4. Epub 2025 Aug 21. PMID 40839334
- [Derived] Hosoya T, Fushimi M, Okui D, Sasaki T, Ohashi T. Open-label study of long-term administration of dotinurad in Japanese hyperuricemic patients with or without gout. Clin Exp Nephrol. 2020 Mar;24(Suppl 1):80-91. doi: 10.1007/s10157-019-01831-5. Epub 2019 Dec 26. PMID 31875931